CLINICAL TRIAL: NCT01726972
Title: A Retrospective Review of FloSeal Use in Total Shoulder Arthroplasty
Status: Completed | Type: Observational
Sponsor: Western Orthopaedics Research and Education Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 369439-1
Record Dates: First submitted 2012-11-08; First posted 2012-11-15 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2012-11

CONDITIONS: Total Shoulder Arthroplasty; Glenohumeral Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The proposed study aims to objectively assess 2-year clinical and radiographic results for the rate of glenoid component loosening in total shoulder arthroplasty (TSA). This retrospective radiographic review will provide evidence for equivalence or superiority in curtailing loosening, a known complication in arthroplasty, when a hemostatic agent is utilized in conjunction with cement at the glenoid.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have completed at least 2 years follow-up following their total shoulder replacement
* Patients must have had radiographic imaging obtained at that 2 years

Exclusion Criteria:

* Patients less than 21 years of age
* Patients who have been imprisoned since the time of surgery
* Patients who are mentally impaired

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have previously undergone anatomic total shoulder arthroplasty for the treatment of glenohumeral osteoarthritis.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2012-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Radiographic Loosening | 2 years
  Radiographic loosening is defined by the presence of radiolucent lines at the bone-cement interface at 2 years. Lines are measured as being either not-present, less than 2mm or greater than/equal to 2mm, in addition to implant seating and the radiodensity between the flanges of the central peg.

CONTACTS AND LOCATIONS:
Locations (1):
- Denver, Colorado, United States